CLINICAL TRIAL: NCT03152396
Title: RxIALTA: Pharmacist CVD Intervention for Patients With Inflammatory Arthritis
Brief Title: Pharmacist CVD Intervention for Patients With Inflammatory Arthritis
Acronym: RxIALTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epidemiology Coordinating and Research Centre, Canada (Other)
Responsible Party: Principal Investigator, Andrea Morgan, Research Coordinator, Epidemiology Coordinating and Research Centre, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072858
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Inflammatory Arthritis; Cardiovascular Risk Factor; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: modifiable cardiovascular risk factors; cardiovascular risk factors; blood pressure; LDL-cholesterol; total-cholesterol; HDL-cholesterol; hemoglobin A1C; tobacco cessation; patient satisfaction
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Tobacco Use Cessation; Patient Satisfaction | interventions — Body Height

STUDY DESIGN:
Intervention Model Description: A non-randomized prospective pre-post-intervention design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with inflammatory arthritis (Other): All patients enrolled have a form of inflammatory arthritis and at least one uncontrolled CV risk factor (i.e. blood pressure, LDL-cholesterol, HbA1C, or current tobacco use). Pharmacist will assess each participants CV risk score using the validated RxEACH CV risk calculator. Over the 6 month intervention period, pharmacists will assist patients to modify a contributing risk factor thru treatment recommendations, prescription adaptation, and prescribing where necessary to meet treatment targets.
  Interventions: Other: CV risk assessment and modification of global risk

INTERVENTIONS:
Other: CV risk assessment and modification of global risk — Individualized CV risk assessment using the validated RxEACH CV risk calculator for baseline and subsequent risk assessment. Pharmacists will assist patient's to decrease CV risk over 6 months thru education, medication modification, and monthly follow-up.
  Other Names: prescription adaptation; prescribing medications; ordering lab work (eg. A1C, lipid panel); interpreting lab work (eg. A1C, lipid panel); blood pressure measurement; height and weight measurements; waist circumference measurement

SUMMARY:
Cardiovascular disease (CVD) (disease of the heart and blood vessels) is one of the leading causes of death and disability in Canada today. The majority of CVD cases are caused by factors that can be controlled. These factors include tobacco use, obesity, high blood pressure, high cholesterol, diabetes, and physical inactivity. Such factors are common and not well controlled. Inflammatory arthritis (IA) (Inflammation of the joints and other tissues) is considered another risk factor or CVD. As such, people who have IA and any of the previously mentioned risk factors would be at high risk for developing CVD. Controlling these factors will bring down the risk of having cardiovascular disease and make the quality of the individuals' life better. Pharmacists work with patients and their family doctors to provide cardiovascular care. Having a pharmacist involved in the care process may help patients with IA reduce their CV risk. Pharmacists are easier to reach and may have more opportunities to educate people about medications. This might lead to better prevention and control of cardiovascular diseases.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is one of the leading causes of morbidity and mortality worldwide and in Canada accounting for nearly one third of the total deaths in both instances.1-2 The majority of CVD cases are caused by modifiable risk factors such as tobacco use, obesity, hypertension, hyperlipidemia, diabetes and physical inactivity.3 Inflammatory arthritis, inclusive of rheumatoid arthritis (RA), psoriatic arthritis (PsA), and ankylosing spondylitis (AS), is also recognized as an independent risk factor for CVD.4-7

It has been reported that the risk of myocardial infarction (MI), heart failure (HF) and CV death among patients with IA is 2-3-fold greater than in the general population.8-10 This increased CV risk reflects the combined impact of systemic inflammation, burden of traditional CVD risk factors and impact of certain medications (e.g. steroids, non-steroidal anti-inflammatories [NSAIDs]).5,6 An elevated risk of CVD can be identified early after IA diagnosis, emphasizing the need for early efforts in CV risk screening.11

Despite being recommended by international IA management guidelines,7 CV risk assessment has not been incorporated into clinicians' daily routine.7 Indeed, it has been reported that such assessments generally only exist in larger centers for non-rheumatology patients.12-14 Moreover, Keeling and colleagues reported that most rheumatologists, who are the main care givers for IA patients, conducted suboptimal CV risk assessments. 15 This gap in care for patients with IA is not consistently absorbed by family physicians due to lack of recognition of CV risk in these patients and competing demands of other healthcare needs (e.g. other chronic diseases, cancer, diabetes). 7

Special considerations need to be taken into account when calculating CV risk in patients with IA, as the 'classic' risk engines (such as Framingham16) might underestimate the overall risk,17 since they have not been adequately evaluated in this patient population.18,5 For example, IA patients who might benefit from lipid-lowering agents may be categorized "low risk" when using the Framingham risk engine.17 As such it has been recommended to use a modified Framingham risk engine (multiply the overall risk with 1.5) in patients with IA. 19

CV risk screening and management in patients with IA takes time and effort, but can be performed by other trained health professionals. As such, it has been recommended to utilize a multidisciplinary approach (integration of rheumatology, cardiology and primary care) to support the care of IA patients.6,20-23 Pharmacists are front line, accessible, primary healthcare professionals who see patients more frequently than any other healthcare provider.24 The efficacy of their interventions in managing chronic diseases including osteoarthritis,25, diabetes,7, 26 dyslipidemia,27 hypertension,28,29 heart failure,30 and CVD 31-34 has been well demonstrated in the literature. Pharmacists can systematically identify patients at high risk of CVD,35 improve their medication use,36 and help them achieve their treatment targets.27,28 In addition to clinical outcomes, pharmacist involvement in patient care is associated with improved patient satisfaction and adherence to therapy.28,35,36 This evidence, coupled with their advanced scope of practice, ideally position pharmacists to conduct CV risk screening and management. In addition, Canadian pharmacists have access to practice guidelines for management and prevention of cardiovascular disease in the general population.37 They also have access to the RxEACH CV risk calculator, an interactive CV screening and management tool, which will help them determine CV risk, simply communicate contributing risks to patients, and show patients the impact of modifying their risks. 34

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) who have a physician-diagnosed IA including

  * Rheumatoid arthritis
  * Psoriatic arthritis
  * Ankylosing spondylitis
  * To be eligible for inclusion, all patients must have at least one uncontrolled risk factor (i.e., blood pressure, LDL-cholesterol, HbA1c, or current tobacco use)

Exclusion Criteria:

* Patients will be excluded if they

  * Are unwilling to participate/sign consent form
  * Are unwilling or unable to participate in regular follow-up visits
  * Are pregnant
  * Have uncontrolled IA (i.e., during a disease exacerbation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in CV risk | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator

SECONDARY OUTCOMES:
change in blood pressure | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator
change in LDL-cholesterol | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator
change in total-cholesterol | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator
change in HDL-cholesterol | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator
change in hemoglobin A1C | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator
tobacco cessation | 6 months
  CV risk re-assessment with validated RxEACH CV risk calculator

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, MSc, Principal Investigator — Epidemiology Coordinating and Research Centre, Canada
Locations (1):
- Calgary Co-operative Association Limited, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Hamarneh YN, Marra C, Gniadecki R, Keeling S, Morgan A, Tsuyuki R. RxIALTA: evaluating the effect of a pharmacist-led intervention on CV risk in patients with chronic inflammatory diseases in a community pharmacy setting: a prospective pre-post intervention study. BMJ Open. 2021 Mar 24;11(3):e043612. doi: 10.1136/bmjopen-2020-043612. PMID 33762234